CLINICAL TRIAL: NCT02956837
Title: An Observer-blind Study to Rank Different Formulations of GSK Biologicals' Investigational RSV Vaccine (GSK3003891A) Administered to Healthy Women
Brief Title: A Study to Rank Different Dosages of Antigen of GlaxoSmithKline (GSK) Biologicals' Investigational Respiratory Syncytial Virus (RSV) Vaccine (GSK3003891A), Based on Their Immune Response and Safety, When Administered to Healthy Adult Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 204812; 2016-001135-12 (EudraCT Number)
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Vaccines; Respiratory Syncytial Viruses; Safety; Reactogenicity; Ranking of Formulations; Immunogenicity
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Respiratory Syncytial Virus Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- GSK3003891A vaccine formulation 1 Group (Experimental): Subjects in this group received a single 30 micrograms (µg) dose injection of the investigational GSK3003891A vaccine at Day 0.
  Interventions: Biological: RSV Vaccine (GSK3003891A) formulation 1
- GSK3003891A vaccine formulation 2 Group (Experimental): Subjects in this group received a single 60µg dose injection of the investigational GSK3003891A vaccine at Day 0.
  Interventions: Biological: RSV Vaccine (GSK3003891A) formulation 2
- GSK3003891A vaccine formulation 3 Group (Experimental): Subjects in this group received a single 120µg dose injection of the investigational GSK3003891A vaccine at Day 0.
  Interventions: Biological: RSV Vaccine (GSK3003891A) formulation 3
- Control Group (Placebo Comparator): Subjects in this group received a single placebo injection at Day 0.
  Interventions: Drug: Placebo (Formulation buffer S9b)

INTERVENTIONS:
Biological: RSV Vaccine (GSK3003891A) formulation 1 — Single dose administered intramuscularly at Day 0 in the deltoid region of the non-dominant arm.
  Arms: GSK3003891A vaccine formulation 1 Group
Biological: RSV Vaccine (GSK3003891A) formulation 2 — Single dose administered intramuscularly at Day 0 in the deltoid region of the non-dominant arm.
  Arms: GSK3003891A vaccine formulation 2 Group
Biological: RSV Vaccine (GSK3003891A) formulation 3 — Single dose administered intramuscularly at Day 0 in the deltoid region of the non-dominant arm.
  Arms: GSK3003891A vaccine formulation 3 Group
Drug: Placebo (Formulation buffer S9b) — A single dose of placebo is administered intramuscularly at Day 0 in the deltoid region of the non-dominant arm.
  Arms: Control Group

SUMMARY:
The purpose of this study is to rank different RSV vaccine dosages of antigen (or formulations) based on safety/reactogenicity and immune response data. The formulations eliciting strong immune responses while maintaining an acceptable safety profile will be considered for further evaluation, including in studies vaccinating pregnant women.

DETAILED DESCRIPTION:
The purpose of the RSV F-021 study that will be conducted in an observer-blind manner during Epoch 1 and single blinded during Epoch 2, is to rank the 3 different doses of the non-adjuvanted investigational RSV PreF-vaccine (30, 60 and 120 μg) based on safety/reactogenicity and immunogenicity data up to 1 month post-vaccination (Day 30). Non-pregnant women aged 18-45 years will be randomized in a 1:1:1:1 ratio to receive one of three dose levels (30, 60, 120 μg) of the RSV PreF vaccine or placebo. The doses eliciting strong immune responses while maintaining an acceptable safety profile will be considered for further evaluation, including in studies vaccinating pregnant women. This will allow evaluation of a wider antigen dose range to determine if there is a dose response relationship in terms of antibody response at the higher dose range that was not present at the lower range.

Since in RSV F-021 the 120ug dosage of the PreF-based investigational RSV vaccine will be tested for the first time in humans, appropriate safety monitoring is planned for this study, including pausing enrolment when the first 25% of subjects from each study group have been vaccinated until review of day 7 post-vaccination safety data by an unblinded GSK internal Safety Review Committee (iSRC) has been completed. The enrolment/vaccination of the remaining subjects can only start following the favourable outcome of this iSRC safety review.

In addition to study visits at Day 0, Day 7 and Day 30 to evaluate primary objective of the study, additional study visits are planned at Day 60 and 90 for further investigation of the immunogenicity and safety/reactogenicity profile of the formulations. A follow-up period has been set up in which the subjects will be contacted at Day 180, 270 and 360. During these contacts, the investigator (or delegate) will ask the subject if she has experienced any serious adverse events and/or any AEs leading to study withdrawal since Day 90/last contact (as applicable), as well as if she has become pregnant during the post-vaccination period. The investigator (or delegate) will also ask the subject about concomitant vaccinations/products/medications that she has received since Day 90/last contact (as applicable) and whether the she had a respiratory tract infection that needed medical attention. Contact should be preferably performed via telephone, or alternatively, if phone contact is not possible, through email/other means where the information can be fully collected.

Healthy, non-pregnant women aged 18 - 45 years will be enrolled in this study:

Women aged 18 - 45 years are selected to match the vaccine's target population, i.e. pregnant women, as closely as possible (gender, age).

Non-pregnant women are selected to avoid unnecessarily exposing a vulnerable population (pregnant women and the foetuses/children) to a higher dose of the vaccine that has not previously been studied in non-pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performance of any study specific procedure.
* Non-pregnant female between, and including, 18 and 45 years of age at the time of study vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study

  * Non-childbearing potential is defined as pre-menarche, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * Has practiced adequate contraception for 30 days prior to study vaccination, and
  * Has a negative pregnancy test on the day of study vaccination, and
  * Has agreed to continue adequate contraception up to 90 days after vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines within 30 days prior to study vaccination, or planned use during the study period.
* Concurrently participating in the active phase of another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Chronic administration of immunosuppressants or other immune-modifying drugs, as well as administration of long-acting immune-modifying drugs, within 6 months prior to study vaccination, or planned administration until 90 days post-vaccination. For corticosteroids, this will mean prednisone ≥ 10 mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the study vaccination, or planned administration until 90 days post-vaccination.
* Planned administration/administration of a vaccine not foreseen by the study protocol within the period starting 30 days before and ending 30 days after study vaccination, with the exception of any licensed influenza vaccine which may be administered ≥ 15 days before or after study vaccination.
* Previous experimental vaccination against RSV.
* History of any neurological disorders or seizures.
* Family history of congenital or hereditary immunodeficiency.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* History of or current autoimmune disease
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality as determined by physical examination and/or Medical History.
* Lymphoproliferative disorder or malignancy within previous 5 years.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study vaccine.
* Hypersensitivity to latex.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Current alcohol and/or drug abuse.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥37.5°C for oral, axillary or tympanic route, or ≥ 38.0°C for rectal route.
  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
  * For subjects with acute disease and/or fever at the time of enrolment, Visit 1/Day 0 will be rescheduled within the allowed recruitment period.
* Body mass index (BMI) > 40 kg/m².
* Pregnant or lactating female.
* Planned move to a location that will prohibit participating in the trial until study conclusion.
* Any other condition that the investigator judges may interfere with study procedures or findings.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 406 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2018-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- GSK Investigational Site, Ghent, Belgium
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (2):
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Paris
- Germany (3):
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Goch, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Steff AM, Cadieux-Dion C, de Lannoy G, Prato MK, Czeszak X, Andre B, Ingels DC, Louckx M, Dewe W, Picciolato M, Maleux K, Fissette L, Dieussaert I. Hamster neogenin, a host-cell protein contained in a respiratory syncytial virus candidate vaccine, induces antibody responses in rabbits but not in clinical trial participants. Hum Vaccin Immunother. 2020 Jun 2;16(6):1327-1337. doi: 10.1080/21645515.2019.1693749. Epub 2020 Jan 17. PMID 31951765
- [Derived] Schwarz TF, McPhee RA, Launay O, Leroux-Roels G, Talli J, Picciolato M, Gao F, Cai R, Nguyen TL, Dieussaert I, Miller JM, Schmidt AC. Immunogenicity and Safety of 3 Formulations of a Respiratory Syncytial Virus Candidate Vaccine in Nonpregnant Women: A Phase 2, Randomized Trial. J Infect Dis. 2019 Oct 22;220(11):1816-1825. doi: 10.1093/infdis/jiz395. PMID 31418022

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 406 subjects initially enrolled in the study, 6 subjects had numbers allocated but did not receive any study vaccine dose, hence only 400 subjects were included in the Total Vaccinated Cohort.
Groups:
- GSK3003891A Vaccine Formulation 2 Group: Subjects in this group received a single 60 µg dose injection of the investigational GSK3003891A vaccine at Day 0.
- GSK3003891A Vaccine Formulation 3 Group: Subjects in this group received a single 120 µg dose injection of the investigational GSK3003891A vaccine at Day 0.
Period: Overall Study
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Started | 100 | 99 | 99 | 102
Completed | 100 | 96 | 97 | 99
Not Completed | 0 | 3 | 2 | 3
Not completed — Serious Adverse Events | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 3
Not completed — Lost to Follow-up | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK3003891A Vaccine Formulation 1 Group: Subjects in this group received a single 30µg dose injection of the investigational GSK3003891A vaccine at Day 0.
- Total: Total of all reporting groups
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group | Total
Number analyzed (Participants) | 100 | 99 | 99 | 102 | 400
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.2 (6.7) | 29.1 (7.2) | 29.6 (7.1) | 29.9 (6.9) | 29.7 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 99 | 99 | 102 | 400
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic Ancestry: African Heritage/African American | 1 | 0 | 2 | 1 | 4
  Geographic Ancestry: Asian - Central/South Asian Heritage | 1 | 1 | 0 | 0 | 2
  Geographic Ancestry: Asian - East Asian Heritage | 0 | 0 | 1 | 0 | 1
  Geographic Ancestry: Asian - South East Asian Heritage | 0 | 0 | 0 | 1 | 1
  Geographic Ancestry: White - Arabic/North African Heritage | 0 | 1 | 2 | 1 | 4
  Geographic Ancestry: White - Caucasian/European Heritage | 96 | 97 | 93 | 98 | 384
  Geographic Ancestry: Unspecified | 2 | 0 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Grade 2 and Grade 3 General Adverse Events (AEs) - Solicited and Unsolicited
Description: Assessed solicited general AEs were fatigue, gastrointestinal symptoms [nausea, vomiting, diarrhea and/or abdominal pain], fever and headache. An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.Grade 2 symptoms = occurrence of symptoms discomforting enough to interfere with daily activities. Grade 3 symptoms = symptoms that prevented normal activities. This primary objective focused only on subjects from the investigational GSK3003891A vaccine groups (GSK3003891A vaccine formulation 1 Group, GSK3003891A vaccine formulation 2 Group and GSK3003891A vaccine formulation 3 Group).
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 100 | 99 | 99 | 102
Participants | 32 | 30 | 24 | 27

2. Primary Outcome: Number of Subjects With Grade 2 and Grade 3 Fever
Description: Grade 2 Fever was defined as oral temperature above (>) 38.5 degrees Celsius (°C) to less than or equal to (≤) 39.5°C. Grade 3 Fever was defined as oral temperature > 39.5°C. This primary objective focused only on subjects from the investigational GSK3003891A vaccine groups (GSK3003891A vaccine formulation 1 Group, GSK3003891A vaccine formulation 2 Group and GSK3003891A vaccine formulation 3 Group).
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 100 | 98 | 99 | 102
Participants
  Grade 2 Fever | 0 | 2 | 1 | 0
  Grade 3 Fever | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Subjects With Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Related SAEs = SAEs assessed by the investigator as related to the vaccination. This primary objective focused only on subjects from the investigational GSK3003891A vaccine groups (GSK3003891A vaccine formulation 1 Group, GSK3003891A vaccine formulation 2 Group and GSK3003891A vaccine formulation 3 Group).
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 100 | 99 | 99 | 102
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Neutralizing Antibody Titers Against RSV-A Subtype
Description: RSV-A is one of the two antigenically distinct subgroups of the Respiratory Synctial Virus (RSV). Antibody titers were determined by neutralization assay and presented as geometric mean titers (GMTs), for a seropositivity cut-off value greater than or equal to (≥) 8 ED60 (Estimated Dilution 60). This primary objective focused only on subjects from the investigational GSK3003891A vaccine groups (GSK3003891A vaccine formulation 1 Group, GSK3003891A vaccine formulation 2 Group and GSK3003891A vaccine formulation 3 Group).
Time Frame: At Day 0
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity at Day 30, which included all evaluable subjects who complied with the post-vaccination blood sampling schedule and for whom post-vaccination immunogenicity results were available for this assay at Day 0.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 98 | 95 | 98 | 100
Titers | 228.8 [193.1 to 271.0] | 249.5 [213.9 to 290.9] | 285.7 [244.5 to 333.9] | 247.1 [211.2 to 289.1]

5. Primary Outcome: Neutralizing Antibody Titers Against RSV-A Subtype
Description: RSV-A is one of the two antigenically distinct subgroups of the Respiratory Synctial Virus (RSV). Antibody titers were determined by neutralization assay and presented as geometric mean titers (GMTs), for a seropositivity cut-off value ≥ 8 ED60 (Estimated Dilution 60). This primary objective focused only on subjects from the investigational GSK3003891A vaccine groups (GSK3003891A vaccine formulation 1 Group, GSK3003891A vaccine formulation 2 Group and GSK3003891A vaccine formulation 3 Group).
Time Frame: At Day 30
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity at Day 30, which included all evaluable subjects who complied with the post-vaccination blood sampling schedule and for whom post-vaccination immunogenicity results were available for this assay at Day 30.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- GSK3003891A Vaccine Formulation 2 Group: Subjects in this group received a single 60 micrograms (µg) dose injection of the investigational GSK3003891A vaccine at Day 0.
- GSK3003891A Vaccine Formulation 3 Group: Subjects in this group received a single 120 micrograms (µg) dose injection of the investigational GSK3003891A vaccine at Day 0.
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 98 | 94 | 98 | 100
Titers | 858.2 [724.7 to 1016.3] | 1114.8 [971.9 to 1278.8] | 1245.5 [1070.3 to 1449.2] | 271.6 [228.0 to 323.5]

6. Primary Outcome: Palivizumab Competing Antibody (PCA) Concentrations
Description: PCA concentrations were determined by Enzyme-Linked Immunosorbent Assay (ELISA), presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (µg/mL), for a seropositivity cut-off ≥ 9.6 µg/mL. This primary objective focused only on subjects from the investigational GSK3003891A vaccine groups (GSK3003891A vaccine formulation 1 Group, GSK3003891A vaccine formulation 2 Group and GSK3003891A vaccine formulation 3 Group).
Time Frame: At Day 0
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 98 | 94 | 96 | 100
µg/mL | 5.7 [5.3 to 6.2] | 5.6 [5.2 to 6.1] | 5.8 [5.3 to 6.3] | 6.0 [5.5 to 6.6]

7. Primary Outcome: Pavilizumab Competing Antibody (PCA) Concentrations
Description: as for outcome 6
Time Frame: At Day 30
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 98 | 94 | 98 | 100
µg/mL | 66.8 [59.0 to 75.8] | 81.2 [72.5 to 90.9] | 83.7 [73.5 to 95.5] | 6.1 [5.5 to 6.8]

8. Secondary Outcome: Number of Subjects With Any, Grade 2, Grade 3 and Medically Attended Solicited Local AEs
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 2 pain = painful when limb was moved and that interfered with every day activities.Grade 3 pain = significant pain at rest, pain that prevented normal every day activity. Grade 2 redness/swelling = redness/swelling spreading beyond (>) 50 millimeters (mm) and up to (and including) 100 mm of injection site.Grade 3 redness/swelling = redness/swelling > 100 mm of injection site. Medically attended symptoms = occurrence of symptoms that required medical advice.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 100 | 98 | 99 | 102
Participants
  Any Pain | 52 | 52 | 51 | 11
  Grade 2 Pain | 5 | 5 | 10 | 1
  Grade 3 Pain | 1 | 0 | 1 | 0
  Medically-attended Pain | 0 | 0 | 0 | 0
  Any Redness (mm) | 6 | 10 | 8 | 1
  Grade 2 Redness (mm) | 2 | 2 | 1 | 0
  Grade 3 Redness | 0 | 0 | 0 | 0
  Medically-attended Redness (mm) | 0 | 0 | 0 | 0
  Any Swelling (mm) | 4 | 6 | 7 | 0
  Grade 2 Swelling (mm) | 1 | 0 | 0 | 0
  Grade 3 Swelling (mm) | 0 | 1 | 0 | 0
  Medically-attended Swelling (mm) | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Subjects With Any, Grade 2, Grade 3, Related and Medically Attended Solicited General AEs
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms (which include nausea, vomiting, diarrhoea and/or abdominal pain), headache, fever [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 2 symptoms = occurrence of symptoms discomforting enough to interfere with daily activities. Grade 3 symptoms = symptoms that prevented normal activities.Related = symptom assessed by the investigator as related to the vaccination. Medically attended symptom = occurrence of symptom that required medical advice.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 100 | 98 | 99 | 102
Participants
  Any Fatigue | 47 | 43 | 45 | 42
  Grade 2 Fatigue | 9 | 14 | 8 | 12
  Grade 3 Fatigue | 3 | 3 | 2 | 1
  Related Fatigue | 37 | 29 | 36 | 33
  Medically-attended Fatigue | 0 | 1 | 1 | 0
  Any Gastrointestinal symptoms | 20 | 23 | 14 | 11
  Grade 2 Gastrointestinal symptoms | 4 | 3 | 1 | 1
  Grade 3 Gastrointestinal symptoms | 1 | 2 | 0 | 1
  Related Gastrointestinal symptoms | 13 | 17 | 10 | 7
  Medically-attended Gastrointestinal symptoms | 0 | 0 | 0 | 0
  Any Headache | 47 | 42 | 41 | 37
  Grade 2 Headache | 11 | 11 | 12 | 10
  Grade 3 Headache | 3 | 2 | 1 | 3
  Related Headache | 30 | 27 | 33 | 29
  Medically-attended Headache | 0 | 1 | 1 | 0
  Any Temperature/(Oral) (°C) | 8 | 8 | 6 | 4
  Related Temperature/(Oral) (°C) | 5 | 1 | 6 | 2
  Medically-attended Temperature/(Oral) (°C) | 0 | 3 | 1 | 0

10. Secondary Outcome: Number of Subjects With Any Unsolicited AEs
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 30-day (Days 0-29) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 100 | 99 | 99 | 102
Participants | 55 | 52 | 46 | 49

11. Secondary Outcome: Number of Subjects With Any SAEs
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 0 up to study end, at Day 360
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 100 | 99 | 99 | 102
Participants | 1 | 3 | 2 | 2

12. Secondary Outcome: Number of Subjects With Any Biochemical and Hematological Laboratory Abnormalities
Description: Biochemical parameters assessed included alanine aminotransferase [ALT], aspartate aminotransferase [AST] and creatinine. Hematological parameters assessed included eosinophils, hemoglobin level, lymphocytes, neutrophils, platelet count and White Blood Cells [WBC]. Abnormal laboratory values at Day 7 were Below, Within and Above normal ranges, as compared to the baseline status of the same parameter, at Day 0 (Unknown, Below, Within and Above normal ranges) [e.g. ALT Below - Within = ALT with below normal value at baseline and within normal values at Day 7].
Time Frame: At Day 7
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with available results for each parameter analyzed, at Day 7.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 100 | 98 | 99 | 102
Participants
  ALT, Below: number analyzed (Participants) | 0 | 0 | 0 | 0
  ALT, Within: number analyzed (Participants) | 99 | 97 | 99 | 102
  ALT, Within: Below | 0 | 0 | 0 | 0
  ALT, Within: Within | 99 | 97 | 99 | 102
  ALT, Within: Above | 0 | 0 | 0 | 0
  ALT, Above: number analyzed (Participants) | 1 | 1 | 0 | 0
  ALT, Above: Below | 0 | 0 |  |
  ALT, Above: Within | 1 | 1 |  |
  ALT, Above: Above | 0 | 0 |  |
  AST, Below: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, Within: number analyzed (Participants) | 99 | 97 | 99 | 100
  AST, Within: Below | 0 | 0 | 0 | 0
  AST, Within: Within | 99 | 97 | 98 | 100
  AST, Within: Above | 0 | 0 | 1 | 0
  AST, Above: number analyzed (Participants) | 1 | 1 | 0 | 1
  AST, Above: Below | 0 | 0 |  | 0
  AST, Above: Within | 1 | 1 |  | 1
  AST, Above: Above | 0 | 0 |  | 0
  Creatinine, Below: number analyzed (Participants) | 6 | 5 | 2 | 2
  Creatinine, Below: Below | 2 | 3 | 2 | 0
  Creatinine, Below: Within | 4 | 2 | 0 | 2
  Creatinine, Below: Above | 0 | 0 | 0 | 0
  Creatinine, Within: number analyzed (Participants) | 93 | 92 | 97 | 99
  Creatinine, Within: Below | 1 | 2 | 4 | 0
  Creatinine, Within: Within | 92 | 90 | 93 | 99
  Creatinine, Within: Above | 0 | 0 | 0 | 0
  Creatinine, Above: number analyzed (Participants) | 1 | 1 | 0 | 1
  Creatinine, Above: Below | 0 | 0 |  | 0
  Creatinine, Above: Within | 0 | 1 |  | 0
  Creatinine, Above: Above | 1 | 0 |  | 1
  Eosinophils, Unknown: number analyzed (Participants) | 1 | 1 | 1 | 1
  Eosinophils, Unknown: Below | 0 | 0 | 0 | 0
  Eosinophils, Unknown: Within | 1 | 1 | 1 | 1
  Eosinophils, Unknown: Above | 0 | 0 | 0 | 0
  Eosinophils, Below: number analyzed (Participants) | 12 | 8 | 10 | 8
  Eosinophils, Below: Below | 5 | 5 | 3 | 6
  Eosinophils, Below: Within | 7 | 3 | 7 | 2
  Eosinophils, Below: Above | 0 | 0 | 0 | 0
  Eosinophils, Within: number analyzed (Participants) | 81 | 86 | 83 | 89
  Eosinophils, Within: Below | 3 | 2 | 4 | 5
  Eosinophils, Within: Within | 77 | 84 | 79 | 81
  Eosinophils, Within: Above | 1 | 0 | 0 | 3
  Eosinophils, Above: number analyzed (Participants) | 2 | 0 | 0 | 0
  Eosinophils, Above: Below | 0 |  |  |
  Eosinophils, Above: Within | 1 |  |  |
  Eosinophils, Above: Above | 1 |  |  |
  Hemoglobin, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  Hemoglobin, Unknown: Below | 0 |  |  | 0
  Hemoglobin, Unknown: Within | 1 |  |  | 1
  Hemoglobin, Unknown: Above | 0 |  |  | 0
  Hemoglobin, Below: number analyzed (Participants) | 20 | 11 | 8 | 11
  Hemoglobin, Below: Below | 12 | 7 | 7 | 7
  Hemoglobin, Below: Within | 8 | 4 | 1 | 4
  Hemoglobin, Below: Above | 0 | 0 | 0 | 0
  Hemoglobin, Within: number analyzed (Participants) | 79 | 85 | 91 | 90
  Hemoglobin, Within: Below | 4 | 1 | 7 | 2
  Hemoglobin, Within: Within | 74 | 84 | 84 | 88
  Hemoglobin, Within: Above | 1 | 0 | 0 | 0
  Hemoglobin, Above: number analyzed (Participants) | 0 | 2 | 0 | 0
  Hemoglobin, Above: Below |  | 0 |  |
  Hemoglobin, Above: Within |  | 1 |  |
  Hemoglobin, Above: Above |  | 1 |  |
  Lymphocytes, Unknown: number analyzed (Participants) | 1 | 1 | 1 | 1
  Lymphocytes, Unknown: Below | 0 | 0 | 0 | 0
  Lymphocytes, Unknown: Within | 1 | 1 | 1 | 1
  Lymphocytes, Unknown: Above | 0 | 0 | 0 | 0
  Lymphocytes, Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  Lymphocytes, Below: Below | 0 |  |  | 1
  Lymphocytes, Below: Within | 1 |  |  | 0
  Lymphocytes, Below: Above | 0 |  |  | 0
  Lymphocytes, Within: number analyzed (Participants) | 93 | 93 | 93 | 96
  Lymphocytes, Within: Below | 1 | 0 | 0 | 0
  Lymphocytes, Within: Within | 92 | 93 | 92 | 94
  Lymphocytes, Within: Above | 0 | 0 | 1 | 2
  Lymphocytes, Above: number analyzed (Participants) | 1 | 1 | 0 | 0
  Lymphocytes, Above: Below | 0 | 0 |  |
  Lymphocytes, Above: Within | 1 | 1 |  |
  Lymphocytes, Above: Above | 0 | 0 |  |
  Neutrophils, Unknown: number analyzed (Participants) | 1 | 1 | 1 | 1
  Neutrophils, Unknown: Below | 0 | 0 | 1 | 0
  Neutrophils, Unknown: Within | 1 | 1 | 0 | 1
  Neutrophils, Unknown: Above | 0 | 0 | 0 | 0
  Neutrophils, Below: number analyzed (Participants) | 4 | 1 | 0 | 3
  Neutrophils, Below: Below | 2 | 0 |  | 1
  Neutrophils, Below: Within | 2 | 1 |  | 2
  Neutrophils, Below: Above | 0 | 0 |  | 0
  Neutrophils, Within: number analyzed (Participants) | 91 | 89 | 90 | 93
  Neutrophils, Within: Below | 2 | 6 | 4 | 8
  Neutrophils, Within: Within | 88 | 81 | 86 | 82
  Neutrophils, Within: Above | 1 | 2 | 0 | 3
  Neutrophils, Above: number analyzed (Participants) | 0 | 4 | 3 | 1
  Neutrophils, Above: Below |  | 0 | 0 | 0
  Neutrophils, Above: Within |  | 4 | 3 | 1
  Neutrophils, Above: Above |  | 0 | 0 | 0
  Platelet count, Unknown: number analyzed (Participants) | 2 | 2 | 0 | 1
  Platelet count, Unknown: Below | 0 | 0 |  | 0
  Platelet count, Unknown: Within | 2 | 2 |  | 1
  Platelet count, Unknown: Above | 0 | 0 |  | 0
  Platelet count, Below: number analyzed (Participants) | 0 | 0 | 0 | 0
  Platelet count, Within: number analyzed (Participants) | 95 | 96 | 99 | 100
  Platelet count, Within: Below | 1 | 1 | 0 | 0
  Platelet count, Within: Within | 93 | 95 | 99 | 100
  Platelet count, Within: Above | 1 | 0 | 0 | 0
  Platelet count, Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  Platelet count, Above: Below | 0 |  |  | 0
  Platelet count, Above: Within | 1 |  |  | 1
  Platelet count, Above: Above | 0 |  |  | 0
  WBC, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  WBC, Unknown: Below | 0 |  |  | 0
  WBC, Unknown: Within | 1 |  |  | 1
  WBC, Unknown: Above | 0 |  |  | 0
  WBC, Below: number analyzed (Participants) | 3 | 0 | 1 | 5
  WBC, Below: Below | 2 |  | 0 | 2
  WBC, Below: Within | 1 |  | 1 | 3
  WBC, Below: Above | 0 |  | 0 | 0
  WBC, Within: number analyzed (Participants) | 95 | 93 | 94 | 94
  WBC, Within: Below | 4 | 4 | 1 | 4
  WBC, Within: Within | 90 | 87 | 92 | 87
  WBC, Within: Above | 1 | 2 | 1 | 3
  WBC, Above: number analyzed (Participants) | 0 | 4 | 3 | 1
  WBC, Above: Below |  | 0 | 0 | 0
  WBC, Above: Within |  | 3 | 3 | 1
  WBC, Above: Above |  | 1 | 0 | 0

13. Secondary Outcome: Number of Subjects With Any Biochemical and Hematological Laboratory Abnormalities
Description: Biochemical parameters assessed included alanine aminotransferase [ALT], aspartate aminotransferase [AST] and creatinine. Hematological parameters assessed included eosinophils, hemoglobin level, lymphocytes, neutrophils, platelet count and White Blood Cells [WBC]. Abnormal laboratory values at Day 30 were Below, Within and Above normal ranges, as compared to the baseline values of the same parameter, at Day 0 (Unknown, Below, Within and Above normal ranges) [e.g. ALT Below - Within = ALT with below normal value at baseline and within normal values at Day 30].
Time Frame: At Day 30
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with available results for each parameter analyzed, at Day 30.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 99 | 98 | 99 | 102
Participants
  ALT, Below: number analyzed (Participants) | 0 | 0 | 0 | 0
  ALT, Within: number analyzed (Participants) | 96 | 97 | 99 | 102
  ALT, Within: Below | 0 | 0 | 0 | 0
  ALT, Within: Within | 93 | 97 | 96 | 101
  ALT, Within: Above | 3 | 0 | 3 | 1
  ALT, Above: number analyzed (Participants) | 1 | 1 | 0 | 0
  ALT, Above: Below | 0 | 0 |  |
  ALT, Above: Within | 1 | 0 |  |
  ALT, Above: Above | 0 | 1 |  |
  AST, Below: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, Within: number analyzed (Participants) | 96 | 97 | 99 | 101
  AST, Within: Below | 0 | 0 | 0 | 0
  AST, Within: Within | 94 | 97 | 97 | 100
  AST, Within: Above | 2 | 0 | 2 | 1
  AST, Above: number analyzed (Participants) | 1 | 1 | 0 | 1
  AST, Above: Below | 0 | 0 |  | 0
  AST, Above: Within | 1 | 0 |  | 1
  AST, Above: Above | 0 | 1 |  | 0
  Creatinine, Below: number analyzed (Participants) | 6 | 5 | 2 | 2
  Creatinine, Below: Below | 1 | 2 | 2 | 2
  Creatinine, Below: Within | 5 | 3 | 0 | 0
  Creatinine, Below: Above | 0 | 0 | 0 | 0
  Creatinine, Within: number analyzed (Participants) | 90 | 92 | 97 | 99
  Creatinine, Within: Below | 1 | 0 | 3 | 2
  Creatinine, Within: Within | 89 | 91 | 93 | 97
  Creatinine, Within: Above | 0 | 1 | 1 | 0
  Creatinine, Above: number analyzed (Participants) | 1 | 1 | 0 | 1
  Creatinine, Above: Below | 0 | 0 |  | 0
  Creatinine, Above: Within | 1 | 0 |  | 1
  Creatinine, Above: Above | 0 | 1 |  | 0
  Eosinophils, Unknown: number analyzed (Participants) | 1 | 1 | 1 | 1
  Eosinophils, Unknown: Below | 0 | 1 | 0 | 0
  Eosinophils, Unknown: Within | 1 | 0 | 1 | 1
  Eosinophils, Unknown: Above | 0 | 0 | 0 | 0
  Eosinophils, Below: number analyzed (Participants) | 12 | 8 | 11 | 8
  Eosinophils, Below: Below | 5 | 4 | 4 | 4
  Eosinophils, Below: Within | 7 | 4 | 7 | 4
  Eosinophils, Below: Above | 0 | 0 | 0 | 0
  Eosinophils, Within: number analyzed (Participants) | 84 | 88 | 86 | 90
  Eosinophils, Within: Below | 3 | 6 | 8 | 7
  Eosinophils, Within: Within | 80 | 82 | 75 | 83
  Eosinophils, Within: Above | 1 | 0 | 3 | 0
  Eosinophils, Above: number analyzed (Participants) | 2 | 0 | 0 | 0
  Eosinophils, Above: Below | 0 |  |  |
  Eosinophils, Above: Within | 1 |  |  |
  Eosinophils, Above: Above | 1 |  |  |
  Hemoglobin, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  Hemoglobin, Unknown: Below | 0 |  |  | 0
  Hemoglobin, Unknown: Within | 1 |  |  | 1
  Hemoglobin, Unknown: Above | 0 |  |  | 0
  Hemoglobin, Below: number analyzed (Participants) | 20 | 11 | 8 | 11
  Hemoglobin, Below: Below | 13 | 6 | 6 | 7
  Hemoglobin, Below: Within | 7 | 5 | 2 | 4
  Hemoglobin, Below: Above | 0 | 0 | 0 | 0
  Hemoglobin, Within: number analyzed (Participants) | 78 | 84 | 91 | 90
  Hemoglobin, Within: Below | 2 | 4 | 5 | 3
  Hemoglobin, Within: Within | 76 | 79 | 86 | 87
  Hemoglobin, Within: Above | 0 | 1 | 0 | 0
  Hemoglobin, Above: number analyzed (Participants) | 0 | 2 | 0 | 0
  Hemoglobin, Above: Below |  | 0 |  |
  Hemoglobin, Above: Within |  | 1 |  |
  Hemoglobin, Above: Above |  | 1 |  |
  Lymphocytes, Unknown: number analyzed (Participants) | 1 | 1 | 1 | 1
  Lymphocytes, Unknown: Below | 0 | 0 | 0 | 0
  Lymphocytes, Unknown: Within | 1 | 1 | 1 | 1
  Lymphocytes, Unknown: Above | 0 | 0 | 0 | 0
  Lymphocytes, Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  Lymphocytes, Below: Below | 0 |  |  | 1
  Lymphocytes, Below: Within | 1 |  |  | 0
  Lymphocytes, Below: Above | 0 |  |  | 0
  Lymphocytes, Within: number analyzed (Participants) | 96 | 95 | 97 | 97
  Lymphocytes, Within: Below | 1 | 0 | 0 | 0
  Lymphocytes, Within: Within | 94 | 94 | 97 | 95
  Lymphocytes, Within: Above | 1 | 1 | 0 | 2
  Lymphocytes, Above: number analyzed (Participants) | 1 | 1 | 0 | 0
  Lymphocytes, Above: Below | 0 | 0 |  |
  Lymphocytes, Above: Within | 1 | 1 |  |
  Lymphocytes, Above: Above | 0 | 0 |  |
  Neutrophils, Unknown: number analyzed (Participants) | 1 | 1 | 1 | 1
  Neutrophils, Unknown: Below | 0 | 0 | 0 | 0
  Neutrophils, Unknown: Within | 1 | 1 | 1 | 1
  Neutrophils, Unknown: Above | 0 | 0 | 0 | 0
  Neutrophils, Below: number analyzed (Participants) | 4 | 1 | 0 | 3
  Neutrophils, Below: Below | 1 | 0 |  | 0
  Neutrophils, Below: Within | 3 | 1 |  | 3
  Neutrophils, Below: Above | 0 | 0 |  | 0
  Neutrophils, Within: number analyzed (Participants) | 94 | 91 | 94 | 94
  Neutrophils, Within: Below | 4 | 1 | 1 | 3
  Neutrophils, Within: Within | 88 | 88 | 92 | 88
  Neutrophils, Within: Above | 2 | 2 | 1 | 3
  Neutrophils, Above: number analyzed (Participants) | 0 | 4 | 3 | 1
  Neutrophils, Above: Below |  | 0 | 0 | 0
  Neutrophils, Above: Within |  | 3 | 3 | 1
  Neutrophils, Above: Above |  | 1 | 0 | 0
  Platelet count, Unknown: number analyzed (Participants) | 2 | 2 | 0 | 1
  Platelet count, Unknown: Below | 0 | 0 |  | 0
  Platelet count, Unknown: Within | 2 | 2 |  | 1
  Platelet count, Unknown: Above | 0 | 0 |  | 0
  Platelet count, Below: number analyzed (Participants) | 0 | 0 | 0 | 0
  Platelet count, Within: number analyzed (Participants) | 94 | 95 | 99 | 100
  Platelet count, Within: Below | 0 | 0 | 0 | 0
  Platelet count, Within: Within | 92 | 94 | 99 | 99
  Platelet count, Within: Above | 2 | 1 | 0 | 1
  Platelet count, Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  Platelet count, Above: Below | 0 |  |  | 0
  Platelet count, Above: Within | 1 |  |  | 1
  Platelet count, Above: Above | 0 |  |  | 0
  WBC, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  WBC, Unknown: Below | 0 |  |  | 0
  WBC, Unknown: Within | 1 |  |  | 1
  WBC, Unknown: Above | 0 |  |  | 0
  WBC, Below: number analyzed (Participants) | 3 | 0 | 2 | 4
  WBC, Below: Below | 2 |  | 1 | 0
  WBC, Below: Within | 1 |  | 1 | 4
  WBC, Below: Above | 0 |  | 0 | 0
  WBC, Within: number analyzed (Participants) | 95 | 93 | 94 | 95
  WBC, Within: Below | 3 | 1 | 3 | 0
  WBC, Within: Within | 90 | 89 | 90 | 90
  WBC, Within: Above | 2 | 3 | 1 | 5
  WBC, Above: number analyzed (Participants) | 0 | 4 | 3 | 1
  WBC, Above: Below |  | 0 | 0 | 0
  WBC, Above: Within |  | 2 | 2 | 1
  WBC, Above: Above |  | 2 | 1 | 0

14. Secondary Outcome: Number of Subjects With Any Biochemical and Hematological Laboratory Abnormalities
Description: Biochemical parameters assessed included alanine aminotransferase [ALT], aspartate aminotransferase [AST] and creatinine. Hematological parameters assessed included eosinophils, hemoglobin level, lymphocytes, neutrophils, platelet count and White Blood Cells [WBC]. Abnormal laboratory values at Day 60 were Below, Within and Above normal ranges, as compared to the baseline status of the same parameter, at Day 0 (Unknown, Below, Within and Above normal ranges) [e.g. ALT Below - Within = ALT with below normal value at baseline and within normal values at Day 60].
Time Frame: At Day 60
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with available results for each parameter analyzed, at Day 60.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 100 | 96 | 98 | 101
Participants
  ALT, Below: number analyzed (Participants) | 0 | 0 | 0 | 0
  ALT, Within: number analyzed (Participants) | 98 | 95 | 98 | 101
  ALT, Within: Below | 0 | 0 | 0 | 0
  ALT, Within: Within | 98 | 95 | 98 | 101
  ALT, Within: Above | 0 | 0 | 0 | 0
  ALT, Above: number analyzed (Participants) | 1 | 1 | 0 | 0
  ALT, Above: Below | 0 | 0 |  |
  ALT, Above: Within | 1 | 1 |  |
  ALT, Above: Above | 0 | 0 |  |
  AST, Below: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, Within: number analyzed (Participants) | 98 | 95 | 98 | 100
  AST, Within: Below | 0 | 0 | 0 | 0
  AST, Within: Within | 98 | 95 | 97 | 100
  AST, Within: Above | 0 | 0 | 1 | 0
  AST, Above: number analyzed (Participants) | 1 | 1 | 0 | 1
  AST, Above: Below | 0 | 0 |  | 0
  AST, Above: Within | 1 | 1 |  | 1
  AST, Above: Above | 0 | 0 |  | 0
  Creatinine, Below: number analyzed (Participants) | 6 | 5 | 2 | 2
  Creatinine, Below: Below | 0 | 3 | 2 | 2
  Creatinine, Below: Within | 6 | 2 | 0 | 0
  Creatinine, Below: Above | 0 | 0 | 0 | 0
  Creatinine, Within: number analyzed (Participants) | 92 | 90 | 96 | 98
  Creatinine, Within: Below | 2 | 3 | 3 | 6
  Creatinine, Within: Within | 89 | 87 | 93 | 91
  Creatinine, Within: Above | 1 | 0 | 0 | 1
  Creatinine, Above: number analyzed (Participants) | 1 | 1 | 0 | 1
  Creatinine, Above: Below | 0 | 0 |  | 0
  Creatinine, Above: Within | 1 | 1 |  | 1
  Creatinine, Above: Above | 0 | 0 |  | 0
  Eosinophils, Unknown: number analyzed (Participants) | 1 | 0 | 1 | 1
  Eosinophils, Unknown: Below | 0 |  | 0 | 0
  Eosinophils, Unknown: Within | 1 |  | 1 | 1
  Eosinophils, Unknown: Above | 0 |  | 0 | 0
  Eosinophils, Below: number analyzed (Participants) | 12 | 8 | 10 | 9
  Eosinophils, Below: Below | 5 | 2 | 4 | 5
  Eosinophils, Below: Within | 7 | 6 | 6 | 4
  Eosinophils, Below: Above | 0 | 0 | 0 | 0
  Eosinophils, Within: number analyzed (Participants) | 85 | 87 | 85 | 91
  Eosinophils, Within: Below | 6 | 4 | 5 | 7
  Eosinophils, Within: Within | 77 | 82 | 77 | 81
  Eosinophils, Within: Above | 2 | 1 | 3 | 3
  Eosinophils, Above: number analyzed (Participants) | 2 | 0 | 0 | 0
  Eosinophils, Above: Below | 0 |  |  |
  Eosinophils, Above: Within | 0 |  |  |
  Eosinophils, Above: Above | 2 |  |  |
  Hemoglobin, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  Hemoglobin, Unknown: Below | 0 |  |  | 0
  Hemoglobin, Unknown: Within | 1 |  |  | 1
  Hemoglobin, Unknown: Above | 0 |  |  | 0
  Hemoglobin, Below: number analyzed (Participants) | 20 | 11 | 8 | 11
  Hemoglobin, Below: Below | 13 | 6 | 5 | 8
  Hemoglobin, Below: Within | 7 | 5 | 3 | 3
  Hemoglobin, Below: Above | 0 | 0 | 0 | 0
  Hemoglobin, Within: number analyzed (Participants) | 79 | 82 | 90 | 89
  Hemoglobin, Within: Below | 5 | 4 | 6 | 7
  Hemoglobin, Within: Within | 74 | 78 | 84 | 81
  Hemoglobin, Within: Above | 0 | 0 | 0 | 1
  Hemoglobin, Above: number analyzed (Participants) | 0 | 2 | 0 | 0
  Hemoglobin, Above: Below |  | 0 |  |
  Hemoglobin, Above: Within |  | 1 |  |
  Hemoglobin, Above: Above |  | 1 |  |
  Lymphocytes, Unknown: number analyzed (Participants) | 1 | 0 | 1 | 1
  Lymphocytes, Unknown: Below | 0 |  | 0 | 0
  Lymphocytes, Unknown: Within | 1 |  | 1 | 1
  Lymphocytes, Unknown: Above | 0 |  | 0 | 0
  Lymphocytes, Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  Lymphocytes, Below: Below | 0 |  |  | 0
  Lymphocytes, Below: Within | 1 |  |  | 1
  Lymphocytes, Below: Above | 0 |  |  | 0
  Lymphocytes, Within: number analyzed (Participants) | 97 | 94 | 95 | 99
  Lymphocytes, Within: Below | 1 | 0 | 1 | 0
  Lymphocytes, Within: Within | 96 | 94 | 93 | 96
  Lymphocytes, Within: Above | 0 | 0 | 1 | 3
  Lymphocytes, Above: number analyzed (Participants) | 1 | 1 | 0 | 0
  Lymphocytes, Above: Below | 0 | 0 |  |
  Lymphocytes, Above: Within | 1 | 1 |  |
  Lymphocytes, Above: Above | 0 | 0 |  |
  Neutrophils, Unknown: number analyzed (Participants) | 1 | 0 | 1 | 1
  Neutrophils, Unknown: Below | 0 |  | 0 | 0
  Neutrophils, Unknown: Within | 1 |  | 1 | 1
  Neutrophils, Unknown: Above | 0 |  | 0 | 0
  Neutrophils, Below: number analyzed (Participants) | 4 | 1 | 0 | 3
  Neutrophils, Below: Below | 0 | 0 |  | 1
  Neutrophils, Below: Within | 4 | 1 |  | 2
  Neutrophils, Below: Above | 0 | 0 |  | 0
  Neutrophils, Within: number analyzed (Participants) | 95 | 90 | 92 | 96
  Neutrophils, Within: Below | 4 | 4 | 4 | 4
  Neutrophils, Within: Within | 89 | 84 | 88 | 89
  Neutrophils, Within: Above | 2 | 2 | 0 | 3
  Neutrophils, Above: number analyzed (Participants) | 0 | 4 | 3 | 1
  Neutrophils, Above: Below |  | 0 | 0 | 0
  Neutrophils, Above: Within |  | 4 | 3 | 1
  Neutrophils, Above: Above |  | 0 | 0 | 0
  Platelet count, Unknown: number analyzed (Participants) | 2 | 2 | 0 | 1
  Platelet count, Unknown: Below | 0 | 0 |  | 0
  Platelet count, Unknown: Within | 2 | 2 |  | 1
  Platelet count, Unknown: Above | 0 | 0 |  | 0
  Platelet count, Below: number analyzed (Participants) | 0 | 0 | 0 | 0
  Platelet count, Within: number analyzed (Participants) | 94 | 93 | 98 | 99
  Platelet count, Within: Below | 0 | 0 | 1 | 0
  Platelet count, Within: Within | 93 | 92 | 97 | 98
  Platelet count, Within: Above | 1 | 1 | 0 | 1
  Platelet count, Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  Platelet count, Above: Below | 0 |  |  | 0
  Platelet count, Above: Within | 1 |  |  | 1
  Platelet count, Above: Above | 0 |  |  | 0
  WBC, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  WBC, Unknown: Below | 0 |  |  | 0
  WBC, Unknown: Within | 1 |  |  | 1
  WBC, Unknown: Above | 0 |  |  | 0
  WBC, Below: number analyzed (Participants) | 3 | 0 | 2 | 5
  WBC, Below: Below | 1 |  | 2 | 3
  WBC, Below: Within | 2 |  | 0 | 2
  WBC, Below: Above | 0 |  | 0 | 0
  WBC, Within: number analyzed (Participants) | 96 | 91 | 93 | 94
  WBC, Within: Below | 2 | 1 | 2 | 1
  WBC, Within: Within | 92 | 86 | 90 | 87
  WBC, Within: Above | 2 | 4 | 1 | 6
  WBC, Above: number analyzed (Participants) | 0 | 4 | 3 | 1
  WBC, Above: Below |  | 0 | 0 | 0
  WBC, Above: Within |  | 3 | 2 | 1
  WBC, Above: Above |  | 1 | 1 | 0

15. Secondary Outcome: Number of Subjects With Any Biochemical and Hematological Laboratory Abnormalities
Description: Biochemical parameters assessed included alanine aminotransferase [ALT], aspartate aminotransferase [AST] and creatinine. Hematological parameters assessed included eosinophils, hemoglobin level, lymphocytes, neutrophils, platelet count and White Blood Cells [WBC]. Abnormal laboratory values at Day 90 were Below, Within and Above normal ranges, as compared to the baseline status of the same parameter, at Day 0 (Unknown, Below, Within and Above normal ranges) [e.g. ALT Below - Within = ALT with below normal value at baseline and within normal values at Day 90].
Time Frame: At Day 90
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with available results for each parameter analyzed, at Day 90.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 100 | 97 | 97 | 99
Participants
  ALT, Below: number analyzed (Participants) | 0 | 0 | 0 | 0
  ALT, Within: number analyzed (Participants) | 99 | 95 | 97 | 99
  ALT, Within: Below | 0 | 0 | 0 | 0
  ALT, Within: Within | 98 | 95 | 97 | 99
  ALT, Within: Above | 1 | 0 | 0 | 0
  ALT, Above: number analyzed (Participants) | 1 | 1 | 0 | 0
  ALT, Above: Below | 0 | 0 |  |
  ALT, Above: Within | 1 | 1 |  |
  ALT, Above: Above | 0 | 0 |  |
  AST, Below: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, Within: number analyzed (Participants) | 99 | 95 | 97 | 98
  AST, Within: Below | 0 | 0 | 0 | 0
  AST, Within: Within | 99 | 95 | 97 | 98
  AST, Within: Above | 0 | 0 | 0 | 0
  AST, Above: number analyzed (Participants) | 1 | 1 | 0 | 1
  AST, Above: Below | 0 | 0 |  | 0
  AST, Above: Within | 1 | 1 |  | 1
  AST, Above: Above | 0 | 0 |  | 0
  Creatinine, Below: number analyzed (Participants) | 6 | 5 | 2 | 2
  Creatinine, Below: Below | 1 | 2 | 2 | 2
  Creatinine, Below: Within | 5 | 3 | 0 | 0
  Creatinine, Below: Above | 0 | 0 | 0 | 0
  Creatinine, Within: number analyzed (Participants) | 93 | 90 | 95 | 96
  Creatinine, Within: Below | 3 | 2 | 4 | 3
  Creatinine, Within: Within | 90 | 88 | 91 | 92
  Creatinine, Within: Above | 0 | 0 | 0 | 1
  Creatinine, Above: number analyzed (Participants) | 1 | 1 | 0 | 1
  Creatinine, Above: Below | 0 | 0 |  | 0
  Creatinine, Above: Within | 1 | 0 |  | 1
  Creatinine, Above: Above | 0 | 1 |  | 0
  Eosinophils, Unknown: number analyzed (Participants) | 1 | 1 | 1 | 1
  Eosinophils, Unknown: Below | 0 | 0 | 0 | 0
  Eosinophils, Unknown: Within | 1 | 1 | 1 | 1
  Eosinophils, Unknown: Above | 0 | 0 | 0 | 0
  Eosinophils, Below: number analyzed (Participants) | 12 | 8 | 11 | 9
  Eosinophils, Below: Below | 6 | 2 | 4 | 4
  Eosinophils, Below: Within | 6 | 6 | 7 | 5
  Eosinophils, Below: Above | 0 | 0 | 0 | 0
  Eosinophils, Within: number analyzed (Participants) | 84 | 87 | 80 | 89
  Eosinophils, Within: Below | 6 | 5 | 8 | 9
  Eosinophils, Within: Within | 76 | 81 | 70 | 80
  Eosinophils, Within: Above | 2 | 1 | 2 | 0
  Eosinophils, Above: number analyzed (Participants) | 2 | 0 | 0 | 0
  Eosinophils, Above: Below | 0 |  |  |
  Eosinophils, Above: Within | 2 |  |  |
  Eosinophils, Above: Above | 0 |  |  |
  Hemoglobin, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  Hemoglobin, Unknown: Below | 0 |  |  | 0
  Hemoglobin, Unknown: Within | 1 |  |  | 1
  Hemoglobin, Unknown: Above | 0 |  |  | 0
  Hemoglobin, Below: number analyzed (Participants) | 20 | 11 | 7 | 11
  Hemoglobin, Below: Below | 11 | 5 | 6 | 7
  Hemoglobin, Below: Within | 9 | 6 | 1 | 4
  Hemoglobin, Below: Above | 0 | 0 | 0 | 0
  Hemoglobin, Within: number analyzed (Participants) | 79 | 84 | 89 | 87
  Hemoglobin, Within: Below | 4 | 3 | 4 | 5
  Hemoglobin, Within: Within | 75 | 81 | 84 | 82
  Hemoglobin, Within: Above | 0 | 0 | 1 | 0
  Hemoglobin, Above: number analyzed (Participants) | 0 | 2 | 0 | 0
  Hemoglobin, Above: Below |  | 0 |  |
  Hemoglobin, Above: Within |  | 1 |  |
  Hemoglobin, Above: Above |  | 1 |  |
  Lymphocytes, Unknown: number analyzed (Participants) | 1 | 1 | 1 | 1
  Lymphocytes, Unknown: Below | 0 | 0 | 0 | 0
  Lymphocytes, Unknown: Within | 1 | 1 | 1 | 1
  Lymphocytes, Unknown: Above | 0 | 0 | 0 | 0
  Lymphocytes, Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  Lymphocytes, Below: Below | 0 |  |  | 1
  Lymphocytes, Below: Within | 1 |  |  | 0
  Lymphocytes, Below: Above | 0 |  |  | 0
  Lymphocytes, Within: number analyzed (Participants) | 96 | 94 | 91 | 97
  Lymphocytes, Within: Below | 1 | 0 | 1 | 1
  Lymphocytes, Within: Within | 95 | 93 | 90 | 95
  Lymphocytes, Within: Above | 0 | 1 | 0 | 1
  Lymphocytes, Above: number analyzed (Participants) | 1 | 1 | 0 | 0
  Lymphocytes, Above: Below | 0 | 0 |  |
  Lymphocytes, Above: Within | 1 | 0 |  |
  Lymphocytes, Above: Above | 0 | 1 |  |
  Neutrophils, Unknown: number analyzed (Participants) | 1 | 1 | 1 | 1
  Neutrophils, Unknown: Below | 0 | 0 | 0 | 0
  Neutrophils, Unknown: Within | 1 | 1 | 1 | 1
  Neutrophils, Unknown: Above | 0 | 0 | 0 | 0
  Neutrophils, Below: number analyzed (Participants) | 4 | 1 | 0 | 3
  Neutrophils, Below: Below | 2 | 0 |  | 1
  Neutrophils, Below: Within | 2 | 1 |  | 2
  Neutrophils, Below: Above | 0 | 0 |  | 0
  Neutrophils, Within: number analyzed (Participants) | 94 | 90 | 88 | 94
  Neutrophils, Within: Below | 3 | 5 | 2 | 1
  Neutrophils, Within: Within | 89 | 83 | 86 | 91
  Neutrophils, Within: Above | 2 | 2 | 0 | 2
  Neutrophils, Above: number analyzed (Participants) | 0 | 4 | 3 | 1
  Neutrophils, Above: Below |  | 0 | 0 | 0
  Neutrophils, Above: Within |  | 4 | 3 | 0
  Neutrophils, Above: Above |  | 0 | 0 | 1
  Platelet count, Unknown: number analyzed (Participants) | 3 | 2 | 0 | 1
  Platelet count, Unknown: Below | 1 | 0 |  | 0
  Platelet count, Unknown: Within | 2 | 2 |  | 1
  Platelet count, Unknown: Above | 0 | 0 |  | 0
  Platelet count, Below: number analyzed (Participants) | 0 | 0 | 0 | 0
  Platelet count, Within: number analyzed (Participants) | 94 | 94 | 96 | 95
  Platelet count, Within: Below | 0 | 1 | 0 | 0
  Platelet count, Within: Within | 91 | 91 | 95 | 95
  Platelet count, Within: Above | 3 | 2 | 1 | 0
  Platelet count, Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  Platelet count, Above: Below | 0 |  |  | 0
  Platelet count, Above: Within | 1 |  |  | 1
  Platelet count, Above: Above | 0 |  |  | 0
  WBC, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  WBC, Unknown: Below | 0 |  |  | 0
  WBC, Unknown: Within | 1 |  |  | 1
  WBC, Unknown: Above | 0 |  |  | 0
  WBC, Below: number analyzed (Participants) | 3 | 0 | 2 | 5
  WBC, Below: Below | 1 |  | 1 | 1
  WBC, Below: Within | 2 |  | 1 | 4
  WBC, Below: Above | 0 |  | 0 | 0
  WBC, Within: number analyzed (Participants) | 96 | 93 | 91 | 92
  WBC, Within: Below | 2 | 1 | 1 | 0
  WBC, Within: Within | 91 | 89 | 89 | 89
  WBC, Within: Above | 3 | 3 | 1 | 3
  WBC, Above: number analyzed (Participants) | 0 | 4 | 3 | 1
  WBC, Above: Below |  | 0 | 0 | 0
  WBC, Above: Within |  | 3 | 3 | 0
  WBC, Above: Above |  | 1 | 0 | 1

16. Secondary Outcome: Number of Subjects With Any Biochemical and Hematological Laboratory Abnormalities, by Maximum Grading
Description: The biochemical and hematological parameters analyzed were ALT, AST, creatinine, eosinophils increase, hemoglobin decrease, lymphocytes decrease, neutrophils decrease, platelet count decrease, WBC decrease and WBC increase, which were graded by FDA Toxicity Grading Scale. Assessed grades over the Day 7- Day 90 period were Unknown, Grade 0 (=no grade), Grade 1 (=mild), Grade 2 (=moderate), Grade 3 (=severe) and Grade 4 (=potentially life-threatening), as compared to the baseline status of the same parameters, at Day 0 (Unknown, Grade 1, Grade 2, Grade 3) [e.g. ALT Grade 0 - Unknown = ALT Grade 0 at baseline versus Unknown grade from Day 7 up to Day 90].
Time Frame: From Day 7 up to Day 90
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with available results for each parameter analyzed, during the considered period.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 100 | 98 | 99 | 102
Participants
  ALT, Grade 0: number analyzed (Participants) | 99 | 97 | 99 | 102
  ALT, Grade 0: Unknown | 0 | 0 | 0 | 0
  ALT, Grade 0: Grade 0 | 96 | 97 | 96 | 101
  ALT, Grade 0: Grade 1 | 2 | 0 | 3 | 1
  ALT, Grade 0: Grade 2 | 0 | 0 | 0 | 0
  ALT, Grade 0: Grade 3 | 1 | 0 | 0 | 0
  ALT, Grade 0: Grade 4 | 0 | 0 | 0 | 0
  ALT, Grade 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  ALT, Grade 1: Unknown | 0 |  |  |
  ALT, Grade 1: Grade 0 | 1 |  |  |
  ALT, Grade 1: Grade 1 | 0 |  |  |
  ALT, Grade 1: Grade 2 | 0 |  |  |
  ALT, Grade 1: Grade 3 | 0 |  |  |
  ALT, Grade 1: Grade 4 | 0 |  |  |
  ALT, Grade 2: number analyzed (Participants) | 0 | 1 | 0 | 0
  ALT, Grade 2: Unknown |  | 0 |  |
  ALT, Grade 2: Grade 0 |  | 0 |  |
  ALT, Grade 2: Grade 1 |  | 0 |  |
  ALT, Grade 2: Grade 2 |  | 1 |  |
  ALT, Grade 2: Grade 3 |  | 0 |  |
  ALT, Grade 2: Grade 4 |  | 0 |  |
  AST, Grade 0: number analyzed (Participants) | 100 | 97 | 99 | 101
  AST, Grade 0: Unknown | 0 | 0 | 0 | 0
  AST, Grade 0: Grade 0 | 98 | 97 | 97 | 101
  AST, Grade 0: Grade 1 | 0 | 0 | 2 | 0
  AST, Grade 0: Grade 2 | 1 | 0 | 0 | 0
  AST, Grade 0: Grade 3 | 0 | 0 | 0 | 0
  AST, Grade 0: Grade 4 | 1 | 0 | 0 | 0
  AST, Grade 1: number analyzed (Participants) | 0 | 1 | 0 | 1
  AST, Grade 1: Unknown |  | 0 |  | 0
  AST, Grade 1: Grade 0 |  | 0 |  | 1
  AST, Grade 1: Grade 1 |  | 0 |  | 0
  AST, Grade 1: Grade 2 |  | 1 |  | 0
  AST, Grade 1: Grade 3 |  | 0 |  | 0
  AST, Grade 1: Grade 4 |  | 0 |  | 0
  Creatinine, Grade 0: Unknown | 0 | 0 | 0 | 0
  Creatinine, Grade 0: Grade 0 | 100 | 98 | 99 | 102
  Creatinine, Grade 0: Grade 1 | 0 | 0 | 0 | 0
  Creatinine, Grade 0: Grade 2 | 0 | 0 | 0 | 0
  Creatinine, Grade 0: Grade 3 | 0 | 0 | 0 | 0
  Creatinine, Grade 0: Grade 4 | 0 | 0 | 0 | 0
  Eosinophils increase, Unknown: number analyzed (Participants) | 1 | 1 | 1 | 1
  Eosinophils increase, Unknown: Unknown | 0 | 0 | 0 | 0
  Eosinophils increase, Unknown: Grade 0 | 1 | 1 | 1 | 1
  Eosinophils increase, Unknown: Grade 1 | 0 | 0 | 0 | 0
  Eosinophils increase, Unknown: Grade 2 | 0 | 0 | 0 | 0
  Eosinophils increase, Unknown: Grade 3 | 0 | 0 | 0 | 0
  Eosinophils increase, Unknown: Grade 4 | 0 | 0 | 0 | 0
  Eosinophils increase, Grade 0: number analyzed (Participants) | 97 | 97 | 98 | 101
  Eosinophils increase, Grade 0: Unknown | 0 | 0 | 0 | 0
  Eosinophils increase, Grade 0: Grade 0 | 94 | 96 | 95 | 99
  Eosinophils increase, Grade 0: Grade 1 | 3 | 1 | 3 | 2
  Eosinophils increase, Grade 0: Grade 2 | 0 | 0 | 0 | 0
  Eosinophils increase, Grade 0: Grade 3 | 0 | 0 | 0 | 0
  Eosinophils increase, Grade 0: Grade 4 | 0 | 0 | 0 | 0
  Eosinophils increase, Grade 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  Eosinophils increase, Grade 1: Unknown | 0 |  |  |
  Eosinophils increase, Grade 1: Grade 0 | 0 |  |  |
  Eosinophils increase, Grade 1: Grade 1 | 1 |  |  |
  Eosinophils increase, Grade 1: Grade 2 | 0 |  |  |
  Eosinophils increase, Grade 1: Grade 3 | 0 |  |  |
  Eosinophils increase, Grade 1: Grade 4 | 0 |  |  |
  Eosinophils increase, Grade 2: number analyzed (Participants) | 1 | 0 | 0 | 0
  Eosinophils increase, Grade 2: Unknown | 0 |  |  |
  Eosinophils increase, Grade 2: Grade 0 | 0 |  |  |
  Eosinophils increase, Grade 2: Grade 1 | 0 |  |  |
  Eosinophils increase, Grade 2: Grade 2 | 1 |  |  |
  Eosinophils increase, Grade 2: Grade 3 | 0 |  |  |
  Eosinophils increase, Grade 2: Grade 4 | 0 |  |  |
  Hemoglobin decrease, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  Hemoglobin decrease, Unknown: Unknown | 0 |  |  | 0
  Hemoglobin decrease, Unknown: Grade 0 | 1 |  |  | 1
  Hemoglobin decrease, Unknown: Grade 1 | 0 |  |  | 0
  Hemoglobin decrease, Unknown: Grade 2 | 0 |  |  | 0
  Hemoglobin decrease, Unknown: Grade 3 | 0 |  |  | 0
  Hemoglobin decrease, Unknown: Grade 4 | 0 |  |  | 0
  Hemoglobin decrease, Grade 0: number analyzed (Participants) | 78 | 86 | 88 | 88
  Hemoglobin decrease, Grade 0: Unknown | 0 | 0 | 0 | 0
  Hemoglobin decrease, Grade 0: Grade 0 | 61 | 74 | 73 | 74
  Hemoglobin decrease, Grade 0: Grade 1 | 14 | 12 | 15 | 13
  Hemoglobin decrease, Grade 0: Grade 2 | 2 | 0 | 0 | 1
  Hemoglobin decrease, Grade 0: Grade 3 | 1 | 0 | 0 | 0
  Hemoglobin decrease, Grade 0: Grade 4 | 0 | 0 | 0 | 0
  Hemoglobin decrease, Grade 1: number analyzed (Participants) | 19 | 12 | 9 | 12
  Hemoglobin decrease, Grade 1: Unknown | 0 | 0 | 0 | 0
  Hemoglobin decrease, Grade 1: Grade 0 | 3 | 2 | 2 | 0
  Hemoglobin decrease, Grade 1: Grade 1 | 11 | 9 | 5 | 10
  Hemoglobin decrease, Grade 1: Grade 2 | 5 | 1 | 2 | 2
  Hemoglobin decrease, Grade 1: Grade 3 | 0 | 0 | 0 | 0
  Hemoglobin decrease, Grade 1: Grade 4 | 0 | 0 | 0 | 0
  Hemoglobin decrease, Grade 2: number analyzed (Participants) | 1 | 0 | 2 | 1
  Hemoglobin decrease, Grade 2: Unknown | 0 |  | 0 | 0
  Hemoglobin decrease, Grade 2: Grade 0 | 0 |  | 0 | 0
  Hemoglobin decrease, Grade 2: Grade 1 | 0 |  | 1 | 0
  Hemoglobin decrease, Grade 2: Grade 2 | 1 |  | 1 | 1
  Hemoglobin decrease, Grade 2: Grade 3 | 0 |  | 0 | 0
  Hemoglobin decrease, Grade 2: Grade 4 | 0 |  | 0 | 0
  Hemoglobin decrease, Grade 3: number analyzed (Participants) | 1 | 0 | 0 | 0
  Hemoglobin decrease, Grade 3: Unknown | 0 |  |  |
  Hemoglobin decrease, Grade 3: Grade 0 | 0 |  |  |
  Hemoglobin decrease, Grade 3: Grade 1 | 0 |  |  |
  Hemoglobin decrease, Grade 3: Grade 2 | 1 |  |  |
  Hemoglobin decrease, Grade 3: Grade 3 | 0 |  |  |
  Hemoglobin decrease, Grade 3: Grade 4 | 0 |  |  |
  Lymphocytes decrease, Unknown: number analyzed (Participants) | 1 | 1 | 1 | 1
  Lymphocytes decrease, Unknown: Unknown | 0 | 0 | 0 | 0
  Lymphocytes decrease, Unknown: Grade 0 | 1 | 1 | 1 | 1
  Lymphocytes decrease, Unknown: Grade 1 | 0 | 0 | 0 | 0
  Lymphocytes decrease, Unknown: Grade 2 | 0 | 0 | 0 | 0
  Lymphocytes decrease, Unknown: Grade 3 | 0 | 0 | 0 | 0
  Lymphocytes decrease, Unknown: Grade 4 | 0 | 0 | 0 | 0
  Lymphocytes decrease, Grade 0: number analyzed (Participants) | 96 | 97 | 97 | 100
  Lymphocytes decrease, Grade 0: Unknown | 0 | 0 | 0 | 0
  Lymphocytes decrease, Grade 0: Grade 0 | 90 | 97 | 93 | 99
  Lymphocytes decrease, Grade 0: Grade 1 | 5 | 0 | 4 | 1
  Lymphocytes decrease, Grade 0: Grade 2 | 1 | 0 | 0 | 0
  Lymphocytes decrease, Grade 0: Grade 3 | 0 | 0 | 0 | 0
  Lymphocytes decrease, Grade 0: Grade 4 | 0 | 0 | 0 | 0
  Lymphocytes decrease, Grade 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Lymphocytes decrease, Grade 1: Unknown | 0 |  | 0 |
  Lymphocytes decrease, Grade 1: Grade 0 | 1 |  | 1 |
  Lymphocytes decrease, Grade 1: Grade 1 | 1 |  | 0 |
  Lymphocytes decrease, Grade 1: Grade 2 | 0 |  | 0 |
  Lymphocytes decrease, Grade 1: Grade 3 | 0 |  | 0 |
  Lymphocytes decrease, Grade 1: Grade 4 | 0 |  | 0 |
  Lymphocytes decrease, Grade 2: number analyzed (Participants) | 1 | 0 | 0 | 1
  Lymphocytes decrease, Grade 2: Unknown | 0 |  |  | 0
  Lymphocytes decrease, Grade 2: Grade 0 | 0 |  |  | 0
  Lymphocytes decrease, Grade 2: Grade 1 | 1 |  |  | 1
  Lymphocytes decrease, Grade 2: Grade 2 | 0 |  |  | 0
  Lymphocytes decrease, Grade 2: Grade 3 | 0 |  |  | 0
  Lymphocytes decrease, Grade 2: Grade 4 | 0 |  |  | 0
  Neutrophils decrease, Unknown: number analyzed (Participants) | 1 | 1 | 1 | 1
  Neutrophils decrease, Unknown: Unknown | 0 | 0 | 0 | 0
  Neutrophils decrease, Unknown: Grade 0 | 1 | 1 | 0 | 1
  Neutrophils decrease, Unknown: Grade 1 | 0 | 0 | 1 | 0
  Neutrophils decrease, Unknown: Grade 2 | 0 | 0 | 0 | 0
  Neutrophils decrease, Unknown: Grade 3 | 0 | 0 | 0 | 0
  Neutrophils decrease, Unknown: Grade 4 | 0 | 0 | 0 | 0
  Neutrophils decrease, Grade 0: number analyzed (Participants) | 94 | 95 | 95 | 95
  Neutrophils decrease, Grade 0: Unknown | 0 | 0 | 0 | 0
  Neutrophils decrease, Grade 0: Grade 0 | 80 | 70 | 82 | 82
  Neutrophils decrease, Grade 0: Grade 1 | 10 | 20 | 11 | 8
  Neutrophils decrease, Grade 0: Grade 2 | 3 | 5 | 2 | 5
  Neutrophils decrease, Grade 0: Grade 3 | 1 | 0 | 0 | 0
  Neutrophils decrease, Grade 0: Grade 4 | 0 | 0 | 0 | 0
  Neutrophils decrease, Grade 1: number analyzed (Participants) | 2 | 1 | 3 | 4
  Neutrophils decrease, Grade 1: Unknown | 0 | 0 | 0 | 0
  Neutrophils decrease, Grade 1: Grade 0 | 0 | 1 | 3 | 2
  Neutrophils decrease, Grade 1: Grade 1 | 1 | 0 | 0 | 1
  Neutrophils decrease, Grade 1: Grade 2 | 1 | 0 | 0 | 1
  Neutrophils decrease, Grade 1: Grade 3 | 0 | 0 | 0 | 0
  Neutrophils decrease, Grade 1: Grade 4 | 0 | 0 | 0 | 0
  Neutrophils decrease, Grade 2: number analyzed (Participants) | 3 | 1 | 0 | 2
  Neutrophils decrease, Grade 2: Unknown | 0 | 0 |  | 0
  Neutrophils decrease, Grade 2: Grade 0 | 0 | 0 |  | 0
  Neutrophils decrease, Grade 2: Grade 1 | 1 | 1 |  | 1
  Neutrophils decrease, Grade 2: Grade 2 | 2 | 0 |  | 1
  Neutrophils decrease, Grade 2: Grade 3 | 0 | 0 |  | 0
  Neutrophils decrease, Grade 2: Grade 4 | 0 | 0 |  | 0
  Platelet count decrease, Unknown: number analyzed (Participants) | 4 | 2 | 0 | 1
  Platelet count decrease, Unknown: Unknown | 1 | 0 |  | 0
  Platelet count decrease, Unknown: Grade 0 | 2 | 2 |  | 1
  Platelet count decrease, Unknown: Grade 1 | 0 | 0 |  | 0
  Platelet count decrease, Unknown: Grade 2 | 0 | 0 |  | 0
  Platelet count decrease, Unknown: Grade 3 | 1 | 0 |  | 0
  Platelet count decrease, Unknown: Grade 4 | 0 | 0 |  | 0
  Platelet count decrease, Grade 0: number analyzed (Participants) | 96 | 95 | 99 | 101
  Platelet count decrease, Grade 0: Unknown | 0 | 0 | 0 | 0
  Platelet count decrease, Grade 0: Grade 0 | 94 | 94 | 97 | 100
  Platelet count decrease, Grade 0: Grade 1 | 1 | 1 | 1 | 1
  Platelet count decrease, Grade 0: Grade 2 | 1 | 0 | 1 | 0
  Platelet count decrease, Grade 0: Grade 3 | 0 | 0 | 0 | 0
  Platelet count decrease, Grade 0: Grade 4 | 0 | 0 | 0 | 0
  Platelet count decrease, Grade 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Platelet count decrease, Grade 1: Unknown |  | 0 |  |
  Platelet count decrease, Grade 1: Grade 0 |  | 0 |  |
  Platelet count decrease, Grade 1: Grade 1 |  | 1 |  |
  Platelet count decrease, Grade 1: Grade 2 |  | 0 |  |
  Platelet count decrease, Grade 1: Grade 3 |  | 0 |  |
  Platelet count decrease, Grade 1: Grade 4 |  | 0 |  |
  WBC decrease, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  WBC decrease, Unknown: Unknown | 0 |  |  | 0
  WBC decrease, Unknown: Grade 0 | 1 |  |  | 1
  WBC decrease, Unknown: Grade 1 | 0 |  |  | 0
  WBC decrease, Unknown: Grade 2 | 0 |  |  | 0
  WBC decrease, Unknown: Grade 3 | 0 |  |  | 0
  WBC decrease, Unknown: Grade 4 | 0 |  |  | 0
  WBC decrease, Grade 0: number analyzed (Participants) | 98 | 98 | 98 | 98
  WBC decrease, Grade 0: Unknown | 0 | 0 | 0 | 0
  WBC decrease, Grade 0: Grade 0 | 92 | 95 | 94 | 94
  WBC decrease, Grade 0: Grade 1 | 6 | 3 | 4 | 4
  WBC decrease, Grade 0: Grade 2 | 0 | 0 | 0 | 0
  WBC decrease, Grade 0: Grade 3 | 0 | 0 | 0 | 0
  WBC decrease, Grade 0: Grade 4 | 0 | 0 | 0 | 0
  WBC decrease, Grade 1: number analyzed (Participants) | 1 | 0 | 1 | 3
  WBC decrease, Grade 1: Unknown | 0 |  | 0 | 0
  WBC decrease, Grade 1: Grade 0 | 0 |  | 0 | 0
  WBC decrease, Grade 1: Grade 1 | 1 |  | 0 | 3
  WBC decrease, Grade 1: Grade 2 | 0 |  | 1 | 0
  WBC decrease, Grade 1: Grade 3 | 0 |  | 0 | 0
  WBC decrease, Grade 1: Grade 4 | 0 |  | 0 | 0
  WBC increase, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  WBC increase, Unknown: Unknown | 0 |  |  | 0
  WBC increase, Unknown: Grade 0 | 1 |  |  | 1
  WBC increase, Unknown: Grade 1 | 0 |  |  | 0
  WBC increase, Unknown: Grade 2 | 0 |  |  | 0
  WBC increase, Unknown: Grade 3 | 0 |  |  | 0
  WBC increase, Unknown: Grade 4 | 0 |  |  | 0
  WBC increase, Grade 0: number analyzed (Participants) | 99 | 94 | 96 | 99
  WBC increase, Grade 0: Unknown | 0 | 0 | 0 | 0
  WBC increase, Grade 0: Grade 0 | 95 | 85 | 91 | 88
  WBC increase, Grade 0: Grade 1 | 3 | 9 | 5 | 11
  WBC increase, Grade 0: Grade 2 | 1 | 0 | 0 | 0
  WBC increase, Grade 0: Grade 3 | 0 | 0 | 0 | 0
  WBC increase, Grade 0: Grade 4 | 0 | 0 | 0 | 0
  WBC increase, Grade 1: number analyzed (Participants) | 0 | 4 | 2 | 2
  WBC increase, Grade 1: Unknown |  | 0 | 0 | 0
  WBC increase, Grade 1: Grade 0 |  | 1 | 1 | 1
  WBC increase, Grade 1: Grade 1 |  | 3 | 1 | 0
  WBC increase, Grade 1: Grade 2 |  | 0 | 0 | 1
  WBC increase, Grade 1: Grade 3 |  | 0 | 0 | 0
  WBC increase, Grade 1: Grade 4 |  | 0 | 0 | 0
  WBC increase, Grade 2: number analyzed (Participants) | 0 | 0 | 1 | 0
  WBC increase, Grade 2: Unknown |  |  | 0 |
  WBC increase, Grade 2: Grade 0 |  |  | 0 |
  WBC increase, Grade 2: Grade 1 |  |  | 1 |
  WBC increase, Grade 2: Grade 2 |  |  | 0 |
  WBC increase, Grade 2: Grade 3 |  |  | 0 |
  WBC increase, Grade 2: Grade 4 |  |  | 0 |

17. Secondary Outcome: Neutralizing Antibody Titers Against RSV-A Subtype
Description: RSV-A is one of the two antigenically distinct subgroups of the Respiratory Synctial Virus (RSV). Antibody titers were determined by neutralization assay and presented as geometric mean titers (GMTs), for a seropositivity cut-off value ≥ 8 ED60.
Time Frame: At Day 60 and Day 90
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity at Day 90, which included all evaluable subjects who complied with the post-vaccination blood sampling schedule and for whom post-vaccination immunogenicity results were available for this assay up to Day 90.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 98 | 92 | 96 | 96
Titers
  Anti-RSV.A, Day 60 | 715.4 [615.8 to 831.1] | 831.9 [733.0 to 944.1] | 965.1 [827.7 to 1125.4] | 311.6 [269.0 to 360.8]
  Anti-RSV.A, Day 90: number analyzed (Participants) | 98 | 92 | 95 | 95
  Anti-RSV.A, Day 90 | 566.5 [494.9 to 648.4] | 732.1 [640.2 to 837.2] | 902.8 [776.4 to 1049.9] | 319.6 [274.2 to 372.4]

18. Secondary Outcome: Neutralizing Antibody Titers Against RSV-B Subtype
Description: RSV-B is one of the two antigenically distinct subgroups of the Respiratory Synctial Virus (RSV). Antibody titers were determined by neutralization assay and presented as geometric mean titers (GMTs), for a seropositivity cut-off value ≥ 6 ED60.
Time Frame: At Day 0, Day 30, Day 60 and Day 90
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 98 | 95 | 98 | 100
Titers
  Anti-RSV.B, Day 0 | 385.6 [318.4 to 466.9] | 392.1 [334.3 to 460.0] | 410.6 [346.5 to 486.5] | 340.2 [289.0 to 400.4]
  Anti-RSV.B, Day 30: number analyzed (Participants) | 98 | 94 | 98 | 100
  Anti-RSV.B, Day 30 | 909.1 [778.5 to 1061.6] | 1004.1 [886.5 to 1137.4] | 1131.7 [987.3 to 1297.2] | 357.7 [309.0 to 414.0]
  Anti-RSV.B, Day 60: number analyzed (Participants) | 98 | 92 | 96 | 96
  Anti-RSV.B, Day 60 | 752.1 [646.7 to 874.6] | 847.1 [746.8 to 960.9] | 923.6 [813.2 to 1048.8] | 409.6 [359.2 to 467.1]
  Anti-RSV.B, Day 90: number analyzed (Participants) | 98 | 92 | 95 | 95
  Anti-RSV.B, Day 90 | 667.8 [572.8 to 778.7] | 804.9 [699.4 to 926.3] | 848.6 [731.4 to 984.7] | 423.2 [359.2 to 498.6]

19. Secondary Outcome: Palivizumab Competing Antibody (PCA) Concentrations
Description: PCA concentrations were determined by Enzyme-Linked Immunosorbent Assay (ELISA), presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (µg/mL), for a seropositivity cut-off value ≥ 9.6 µg/mL.
Time Frame: At Day 60 and Day 90
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 98 | 92 | 96 | 96
µg/mL
  PCA, Day 60 | 55.2 [48.8 to 62.5] | 69.0 [62.4 to 76.4] | 66.7 [58.7 to 75.8] | 6.4 [5.8 to 7.1]
  PCA, Day 90: number analyzed (Participants) | 98 | 92 | 94 | 95
  PCA, Day 90 | 47.6 [42.3 to 53.5] | 57.9 [51.4 to 65.1] | 57.0 [50.0 to 64.9] | 7.4 [6.5 to 8.6]

20. Secondary Outcome: Antibody Concentrations Against Neogenin (NEO) Residual Host Cell Protein
Description: Anti-neogenin (anti-NEO) antibody concentrations were determined by ELISA, presented as geometric mean concentrations (GMCs) and expressed in nanograms per milliliter (ng/mL), for a seropositivity cut-off value ≥ 55 ng/mL.
Time Frame: At Day 0 and Day 30
Population: This immunogenicity analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom immunogenicity results were available for this assay up to Day 30.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 100 | 99 | 99 | 102
ng/mL
  Anti-NEO, Day 0: number analyzed (Participants) | 100 | 99 | 97 | 102
  Anti-NEO, Day 0 | 32.9 [29.2 to 37.1] | 32.0 [28.7 to 35.7] | 33.5 [29.3 to 38.3] | 34.5 [30.0 to 39.5]
  Anti-NEO, Day 30: number analyzed (Participants) | 100 | 98 | 99 | 102
  Anti-NEO, Day 30 | 32.9 [29.5 to 36.7] | 31.5 [28.4 to 34.9] | 33.1 [29.3 to 37.4] | 34.7 [30.2 to 39.9]

21. Secondary Outcome: Number of Subjects With Any Medically Attended (MA) Respiratory Tract Infections (RTIs) Associated With RSV
Description: MA-RSV-RTIs were defined as a visit to a health care provider for respiratory symptoms including but not limited to cough, sputum production, difficulty breathing.
Time Frame: From Day 0 up to study end, at Day 360
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
Number analyzed (Participants) | 100 | 99 | 99 | 102
Participants | 21 | 11 | 10 | 9

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited symptoms: during the 30-day (Days 0-29) post-vaccination period; SAEs: during the entire study period (Day 0-Day 360).
Arm/Group | GSK3003891A Vaccine Formulation 1 Group | GSK3003891A Vaccine Formulation 2 Group | GSK3003891A Vaccine Formulation 3 Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/99 | 0/99 | 0/102
Serious Adverse Events (participants affected / at risk) | 1/100 | 3/99 | 2/99 | 2/102
Other Adverse Events (participants affected / at risk) | 88/100 | 86/99 | 83/99 | 76/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3003891A Vaccine Formulation 1 Group (N=100) | GSK3003891A Vaccine Formulation 2 Group (N=99) | GSK3003891A Vaccine Formulation 3 Group (N=99) | Control Group (N=102)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3003891A Vaccine Formulation 1 Group (N=100) | GSK3003891A Vaccine Formulation 2 Group (N=99) | GSK3003891A Vaccine Formulation 3 Group (N=99) | Control Group (N=102)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 22 (22) | 24 (24) | 14 (14) | 11 (11)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (3) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 47 (48) | 43 (43) | 45 (46) | 42 (42)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Injection site pruritus (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 52 (53) | 52 (52) | 51 (51) | 11 (12)
Pyrexia (General disorders) | 8 (8) | 8 (8) | 6 (6) | 4 (4)
Swelling (General disorders) | 4 (4) | 6 (6) | 7 (7) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 3 (4) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infective keratitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 6 (7) | 3 (3) | 4 (4) | 4 (5)
Oral herpes (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 13 (14) | 3 (4) | 7 (7) | 6 (6)
Salpingo-oophoritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 9 (10) | 8 (8) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3) | 1 (1) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Facial neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 54 (61) | 47 (56) | 47 (55) | 47 (53)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Menstrual disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polymenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Premenstrual pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 5 (5) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 4 (4) | 4 (4) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 6 (6) | 10 (10) | 8 (8) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT02956837/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT02956837/SAP_001.pdf